CLINICAL TRIAL: NCT02871284
Title: Prevention of Chemotherapy-Related Polyneuropathy Via Sensorimotor Exercise Training
Acronym: PIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: University Hospital Heidelberg (Other); National Center for Tumor Diseases, Heidelberg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-630/2015/PIC
Record Dates: First submitted 2016-05-06; First posted 2016-08-18 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Exercise; Chemotherapy-induced Polyneuropathy
Keywords: cancer; anticancer treatment; exercise; physical activity; sensorimotor training; chemotherapy-induced polyneuropathy
MeSH Terms: conditions — Motor Activity; Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sensorimotor training (EI) (Experimental): The participants of the experimental intervention arm will take part in a 45 minutes sensorimotor training class two times a week for a maximum of 24 weeks at the NCT (National Center for Tumor Diseases). Highly qualified exercise therapists will guide the class. Class size will be no bigger than 8 patients to ensure adequate individual supervision and guidance. Additionally, participants will be asked to perform one weekly 15 minutes home-based sessions without supervision. Participants who are not able to come to the NCT Heidelberg 2x/week will be offered a home-based sensorimotor program including the same exercises. At the beginning, participants will receive an appointment for an individual face-to-face counseling session at the NCT. During this appointment, the patient will receive an exercise manual for individualized home-based sensorimotor training and a practical introduction by the exercise therapist.
  Interventions: Behavioral: Exercise
- machine-based resistance training (AC) (Active Comparator): Participants of the active control arm will receive machine-based resistance training. The supervised resistance exercise program will be undertaken twice weekly in small groups (not more than 12 people per group) of participants and will be guided by an exercise physiotherapist over a maximum of 24 weeks. All sessions will start with a warm-up and finish with a cool-down (comprising exercise on a cycle ergometer or treadmill at a relatively low intensity and stretching activities) and will take approximately 45 minutes. Additionally, participants will be asked to perform a weekly 15 minutes home-based resistance training session without supervision
  Interventions: Behavioral: Exercise
- usual care (No Intervention): Participants will receive usual care with no additional exercise training or intervention

INTERVENTIONS:
Behavioral: Exercise
  Arms: Sensorimotor training (EI); machine-based resistance training (AC)

SUMMARY:
Chemotherapy-induced peripheral neurotoxicity (CIPN) as a side effect of chemotherapy negatively affects patients' quality of life and may lead to treatment disturbances. CIPN is frequently recorded in patients treated with alkylating platinum-based drugs, antitubulins including the taxanes and vinca alkaloids, and other drugs including suramin, thalidomide, lenalidomide and the proteasome inhibitor bortezomib, representing one of the most severe and potentially dose-limiting non-hematological toxic effects. Sufficient treatment options or preventive measures are lacking.

There is evidence that physical activity strategies are able to address existing CIPN symptoms and potentially increase quality of life in affected patients. CIPN symptoms involves restrictions of sensory and sometimes motor modalities, for example, deficits in plantar perception and dysfunction of postural control and one study in type II diabetes patients also suggested that structured exercise might have a preventive potential with regard to peripheral neuropathy incidence.

Based on these findings, we aim to investigate the preventive potential of a sensorimotor intervention vs. machine-based resistance training vs. usual care (wait-list control group) in a randomized controlled three-arm intervention trial among cancer patients undergoing chemotherapy with high risk for CIPN. On the basis of power calculations, the goal is to include 82 patients per intervention arm resulting in a total patients number to be enrolled of n=246. CIPN symptoms will be assessed objectively via comprehensive clinical and electrodiagnostic examinations (Total Neuropathy Scale; TNS-reduced) and subjectively via questionnaires (EORTC QLQ-CIPN20 & FACT-GOG-Ntx, EORTC QLQ-C30). Additionally CIPN and the effectiveness of the selected interventions will be objectively evaluated by spectral analysis of Centre of Pressure (COP) variations. Further key secondary endpoints are: physical performance, sleep quality and chemotherapy compliance.

ELIGIBILITY:
Inclusion Criteria:

diagnosed with cancer and assigned to receive a chemotherapeutic regimen containing at least one of the following agents:

* a platinum analog, e.g., cisplatin, carboplatin, oxaliplatin
* a vinca alkaloid, e.g., vincristine
* a taxane, e.g., paclitaxel, docetaxel
* suramin
* thalidomide or lenalidomide
* bortezomib

Physical capability that allows the performance of the training program implemented within the experimental intervention or the control intervention arm

Exclusion Criteria:

* Known polyneuropathy of any kind or any polyneuropathic signs or symptoms at baseline
* Abnormal electroneurographic findings at baseline
* Known metastasis to the central or peripheral nervous system
* Any physical or mental handicap that would hamper the performance of the training program implemented within the intervention arms
* Family history positive for any hereditary polyneuropathy
* Known history of alcohol or illegal drug abuse or any constellation of lab values suggesting alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Total Neuropathy Scale (TNS) | up to week 24 (and 3 & 6 month follow up)
  The TNS is based on symptoms, signs and basic instrumental evaluations and provides a much larger range of scoring values (0 - 40) than common oncological toxicity scales such as the National Cancer Institute (NCI) Common Toxicity Criteria (ranging from 0 - 4, cf. http://ctep.cancer.gov/forms), thus allowing the severity of CIPN to be graded more precisely. The TNS has so far been used to assess the neurotoxicity of various CIPN-relevant chemotherapeutic agents, and its results are clearly correlated with the clinically relevant results of NCI Common Toxicity Criteria, Ajani's and Eastern Cooperative Oncology Group toxicity scales, which are commonly used by oncologists.28-32 Within the PIC-Study the TNS-reduced will the primary endpoint. The TNS-reduced score excludes QST (quantitative sensory testing) vibration testing resulting in a TNS scale from 0-36.

SECONDARY OUTCOMES:
Centre of Pressure (COP) | up to week 24 (and 3 & 6 month follow up)
  total COP displacement; mean velocity (anterior-posterior; medial-lateral) and frequency. This is just one assessement with various outcome variables
Strength Performance | up to week 24
  Isometric (in four different joint angle positions) and isokinetic (at 60° angle speed) muscle capacity is measured with the Isomed 2000® diagnostic module. The protocol includes testing of representative muscles groups for upper (elbow flexors/extensors) and lower extremity (knee extensors/flexors) and is currently well established in different ongoing and finished studies in our unit.
Cardiopulmonary Fitness | up to week 24 (and 3 & 6 month follow up)
  Maximal endurance performance (VO2peak) is measured by performing a maximal bicycle ergometer test (CPET) with a quasi-ramp protocol starting at 20 watts and increasing by 10 watts every minute until volitional exhaustion.
EORTC QLQ-C30 | up to week 24 (and 3 & 6 month follow up)
  QoL will be assessed with the validated 30-item self-assessment questionnaire of the European Organisation for Research and Treatment of Cancer (EORTC QLQ-C30, version 3.0). It includes five multi-item functional scales (physical, role, emotional, cognitive, and social function), three multi-item symptom scales (fatigue, pain, nausea/vomiting), and six single items assessing further symptoms (dyspnea, insomnia, appetite loss, constipation, diarrhea) and financial difficulties.
EORTC QLQ-CIPN20 | prior to each Chemotherapy cycle within the first 24 weeks (and 3 & 6 month follow up)
  The EORTC QLQ-CIPN20 is a 20-item quality of life questionnaire, which has been developed to elicit patients' experience of symptoms and functional limitations related to CIPN. The CIPN20 has three subscales: a sensory, motor, and autonomic subscale. In combination with the more classical, physician-based clinical rating scales, the CIPN20 should yield a more complete picture of the nature, frequency, and severity of CIPN in a wide range of oncology patient populations. This phase IV questionnaire has been field tested in a large international clinical trial and the data are currently being analyzed.
FACT-GOG-Ntx | prior to each Chemotherapy cycle within the first 24 weeks (and 3 & 6 month follow up)
  The FACT-GOG-Ntx is an eleven-item scale that evaluates symptoms and concerns associated specifically with chemotherapy-induced peripheral neuropathy. The questionnaire has been validated, ranges from zero to 44 with higher scores indicating increased CIPN symptoms and has been used in various clinical trials.
Multidimensional Fatigue Inventory (MFI) | up to week 24 (and 3 & 6 month follow up)
  Fatigue will be assessed with the Multidimensional Fatigue Inventory (MFI) which is a 20-item, multidimensional self-assessment questionnaire that has been validated for a German-speaking population. It covers five different dimensions of fatigue (general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue). Scores are derived by summing the answers (five-stage scale) of the appropriate items. The MFI has been used to assess fatigue in a variety of cancer patient studies, and psychometric properties of this instrument have been classified as satisfying or good.
Pittsburgh Sleep Quality Index (PSQI) | up to week 24 (and 3 & 6 month follow up)
  Sleep quality and sleep problems will be assessed with the validated and frequently used Pittsburgh Sleep Quality Index
Short QUestionnaire to ASsess Health-enhancing Physical Activity | up to week 24 (and 3 & 6 month follow up)
  Physical activity behavior (PA) in the domains of commuting activity, leisure time activities such as cycling, walking, and sports, household and occupational activity will be assessed via a standardized and validated questionnaire, the Short QUestionnaire to ASsess Health-enhancing PA (SQUASH) which has the advantage that it is short and easy to complete.

OTHER OUTCOMES:
Safety of exercise interventions | up to week 24
  Physical behavior and well-being will be recorded by the participant (exercise log) prior to and after each training session. Pain, nausea, dyspnea, and other adverse events, in particular those deemed to be causally related to the study interventions, are systematically documented by questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Tumor Diseases, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Pooling Initiative with the STOP Trial

REFERENCES:
- [Derived] Muller J, Weiler M, Schneeweiss A, Haag GM, Steindorf K, Wick W, Wiskemann J. Preventive effect of sensorimotor exercise and resistance training on chemotherapy-induced peripheral neuropathy: a randomised-controlled trial. Br J Cancer. 2021 Sep;125(7):955-965. doi: 10.1038/s41416-021-01471-1. Epub 2021 Jul 5. PMID 34226683